CLINICAL TRIAL: NCT00353678
Title: Direct Factor Xa Inhibitor YM150 for Prevention of Venous Thromboembolism in Patients Undergoing Elective Total Hip Replacement.---A Double Blind, Parallel, Dose-finding Study in Comparison With Open Label Enoxaparin
Brief Title: Factor Xa Inhibitor YM150 for the Prevention of Blood Clot Formation in Veins After Scheduled Hip Replacement (ONYX-2)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 150-CL-008
Record Dates: First submitted 2006-07-18; First posted 2006-07-19 (Estimated); Last update posted 2013-03-21 (Estimated); Status verified 2013-03

CONDITIONS: Thromboembolism
Keywords: Hip replacement; Arthroplasty; Prevention; Thromboembolism; Treatment outcomes; Arthroplasty, replacement, hip
MeSH Terms: conditions — Thromboembolism

INTERVENTIONS:
Drug: YM150

SUMMARY:
The purpose of this study is to find the best possible (optimal) dose (effect versus adverse events) of YM150 to prevent the risk of blood clot formation after scheduled hip replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective primary hip replacement
* Age 18 years or over
* Written informed consent obtained

Exclusion Criteria:

* Documented history or considered at increased risk of venous thromboembolism
* Subjects considered at increased risk of bleeding
* Surgery planned for contralateral hip at the same time or within 10 weeks after enrolment
* Concomitant use of anticoagulants/ antiplatelet agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1141 (Actual)
Dates: Start 2006-06; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Rate of total venous thromboembolism (VTE) during hospitalization phase
Incidence of clinically relevant bleeding during 7-10 days hospitalization treatment rated as Major

SECONDARY OUTCOMES:
Proximal or distal deep vein thrombosis (DVT) during hospitalization phase
Symptomatic VTE
Rate of total VTE
Death due to any cause during treatment
Incidence of the bleeding types:
Major or clinically relevant non-major bleeding, Major bleeding,
Clinically relevant non-major bleeding, Minor bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Astellas Pharma Europe B.V., Medical Clinical Development, Principal Investigator — Department of Orthopedics, Surgical Sciences, Gothenburg University Sahlgrenska/ÖSTRA University Hospital, Goteborg, Sweden
Locations (68):
- Austria (2):
  - Innsbruck
  - Vienna
- Bosnia and Herzegovina (3):
  - Foča
  - Sarajevo
  - Tuzla
- Czechia (4):
  - Brno
  - Kladno
  - Prague
  - Třebíč
- Denmark (4):
  - Copenhagen
  - Herlev
  - Hørsholm
  - Silkeborg
- Finland (2):
  - Jyväskylä
  - Oulu
- Germany (6):
  - Berlin
  - Frankfurt am Main
  - Halle
  - Kremmen OT Somerfeld
  - Markgröningen
  - Schwandorf in Bayern
- Greece (2):
  - Athens
  - Melíssia
- Italy (9):
  - Bologna
  - Milan
  - Parma
  - Pavia
  - Pietra Ligure
  - Reggio Emilia
  - Rozzano
  - S. Donato Milanese
  - Udine
- Latvia (2):
  - Riga
  - Valmiera
- Lithuania (2):
  - Kaunas
  - Vilnius
- Norway (3):
  - Elverum
  - Trondheim
  - Tynset
- Poland (5):
  - Bialystok
  - Katowice
  - Krakow
  - Lublin
  - Warsaw
- Russia (7):
  - Chelyabinsk
  - Moscow
  - Nizhny Novgorod
  - Orenburg
  - Saint Petersburg
  - Samara
  - Volgograd
- Serbia (5):
  - Belgrade
  - Kragujevac
  - Niš
  - Novi Sad
  - Subotica
- Slovakia (2):
  - Banska Bysterica
  - Ružomberok
- Spain (5):
  - Cantoria
  - Castellon
  - Cáceres
  - Madrid
  - Valencia
- Sweden (5):
  - Falköping
  - Gothenburg
  - Kalmar
  - Motala
  - Stockholm

REFERENCES:
- [Background] Eriksson BI, Turpie AG, Lassen MR, Prins MH, Agnelli G, Kalebo P, Wetherill G, Wilpshaar JW, Meems L; ONYX-2 STUDY GROUP. Prevention of venous thromboembolism with an oral factor Xa inhibitor, YM150, after total hip arthroplasty. A dose finding study (ONYX-2). J Thromb Haemost. 2010 Apr;8(4):714-21. doi: 10.1111/j.1538-7836.2010.03748.x. Epub 2010 Jan 17. PMID 20088935